CLINICAL TRIAL: NCT02246218
Title: An Open Label Study of the Safety, Efficacy and Pharmacokinetics of Glycerol Phenylbutyrate (GPB; RAVICTI®) in Pediatric Subjects Under Two Years of Age With Urea Cycle Disorders (UCDs)
Brief Title: A Study of the Safety, Efficacy and Pharmacokinetics of Glycerol Phenylbutyrate in Pediatric Subjects Under 2 Years of Age With Urea Cycle Disorders
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HPN-100-009; 2016-003460-38 (EudraCT Number)
Record Dates: First submitted 2014-09-17; First posted 2014-09-22 (Estimated); Results first posted 2019-03-05 (Actual); Last update posted 2024-07-01 (Actual); Status verified 2024-06

CONDITIONS: Urea Cycle Disorder
Keywords: Urea Cycle Disorder; UCD; Buphenyl; Glycerol Phenylbutyrate; Ravicti; Hyperammonemia; Sodium Phenylbutyrate; GPB; HPN-100
MeSH Terms: conditions — Urea Cycle Disorders, Inborn; Hyperammonemia | interventions — glycerol phenylbutyrate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- RAVICTI (Experimental): RAVICTI Oral Liquid should be administered just prior to breastfeeding or intake of formula or food. The recommended dosing regimen is 3-6 times per day depending on feeding schedule and at the discretion of the Investigator.
  Interventions: Drug: RAVICTI

INTERVENTIONS:
Drug: RAVICTI
  Other Names: HPN-100; Glycerol Phenylbutyrate; GPB

SUMMARY:
This is an open-label study consisting of a transition period to RAVICTI, followed by a safety extension period for at least 6 months and up to 24 months of treatment with RAVICTI, depending on age at enrollment. It is designed to capture information important for evaluating safety, pharmacokinetics and efficacy in young children.

Subjects who are followed by or referred to the Investigator for management of their UCD. Subjects eligible for this study will include patients ranging from newborn to < 2 years of age with either a diagnosed or clinically suspected UCD.

DETAILED DESCRIPTION:
Study acquired from Horizon in 2024.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects up to 2 years of age
* Signed informed consent by subject's parent/legal guardian
* UCD diagnosis or suspected diagnosis of any subtype, except N-acetyl glutamate synthetase deficiency. If UCD has not been previously confirmed by genetic testing, consent must be obtained from parent/legal guardian prior to perform genetic testing. If genetic testing is inconsistent with or excludes a UCD diagnosis, the subject will be withdrawn from the study.

Exclusion Criteria:

* Use of any investigational drug within 30 days of Day 1
* Uncontrolled infection (viral or bacterial) or any other condition known to precipitate hyperammonemic crises. Once these precipitating factors are medically controlled, patients presenting in crisis are eligible.
* Any clinical or laboratory abnormality of Grade 3 or greater severity according to the Common Terminology Criteria for Adverse Events (CTCAE) v4.03, except Grade 3 elevations in ammonia and liver enzymes, defined as levels 5-20 times the upper limit of normal in alanine aminotransferase (ALT), aspartate aminotransferase (AST), or gamma glutamyl transpeptidase (GGT) in a clinically stable subject
* Any clinical or laboratory abnormality or medical condition that, at the discretion of the Investigator, may put the subject at increased risk by participating in this study
* Known hypersensitivity to phenylacetate (PAA) or phenylbutyrate (PBA)
* Liver transplantation, including hepatocellular transplant
* Subjects on hemodialysis at time of initiating RAVICTI
* Subjects on RAVICTI for UCD management
* Currently treated with Carbaglu® (carglumic acid)

Ages: 1 Day to 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 27 (Actual)
Dates: Start 2014-12-31 (Actual); Primary Completion 2016-10-17 (Actual); Study Completion 2017-07-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (17):
- United States (16):
  - Kaiser Permanente Regional Metabolic Center, Los Angeles, California
  - Stanford Center for Clinical & Translational Research & Education, Palo Alto, California
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Shands at University of Florida, Gainesville, Florida
  - Emory University, Decatur, Georgia
  - Indiana University, Indianapolis, Indiana
  - Maine Medical Center, Portland, Maine
  - Children's Hospital of Michigan, Detroit, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Mount Sinai School of Medicine, New York, New York
  - University Hospitals Case Medical Center, Cleveland, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - University of Utah, Salt Lake City, Utah
  - Seattle Children's Hospital, Seattle, Washington
- The Hospital for Sick Children, Toronto, Canada

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: https://www.amgen.com/datasharing

REFERENCES:
- [Result] Berry SA, Longo N, Diaz GA, McCandless SE, Smith WE, Harding CO, Zori R, Ficicioglu C, Lichter-Konecki U, Robinson B, Vockley J. Safety and efficacy of glycerol phenylbutyrate for management of urea cycle disorders in patients aged 2months to 2years. Mol Genet Metab. 2017 Nov;122(3):46-53. doi: 10.1016/j.ymgme.2017.09.002. Epub 2017 Sep 8. PMID 28916119
- [Result] Berry SA, Vockley J, Vinks AA, Dong M, Diaz GA, McCandless SE, Smith WE, Harding CO, Zori R, Ficicioglu C, Lichter-Konecki U, Perdok R, Robinson B, Holt RJ, Longo N. Pharmacokinetics of glycerol phenylbutyrate in pediatric patients 2 months to 2 years of age with urea cycle disorders. Mol Genet Metab. 2018 Nov;125(3):251-257. doi: 10.1016/j.ymgme.2018.09.001. Epub 2018 Sep 4. PMID 30217721
- See also: Related Info — https://www.ravicti.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 27 participants were enrolled; 1 participant was not dosed and is not included in any analysis.
Groups:
- RAVICTI: Age 2 Months to < 2 Years: Participants age 2 months to < 2 years received RAVICTI Oral Liquid administered just prior to breastfeeding or intake of formula or food. The recommended dosing regimen is 3-6 times per day depending on feeding schedule and at the discretion of the Investigator.
- RAVICTI: Age 0 to < 2 Months: Participants age 0 to < 2 months received RAVICTI Oral Liquid administered just prior to breastfeeding or intake of formula or food. The recommended dosing regimen is 3-6 times per day depending on feeding schedule and at the discretion of the Investigator.
Period: Overall Study
Arm/Group | RAVICTI: Age 2 Months to < 2 Years | RAVICTI: Age 0 to < 2 Months
Started | 10 | 16
Completed | 6 | 10
Not Completed | 4 | 6
Not completed — Withdrawal by Parent/Guardian | 0 | 1
Not completed — Stopping Rule: Liver Transplant | 2 | 4
Not completed — Adverse Event | 1 | 1
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- RAVICTI: Age 0 to <2 Months: Participants age 0 to < 2 months received RAVICTI Oral Liquid administered just prior to breastfeeding or intake of formula or food. The recommended dosing regimen is 3-6 times per day depending on feeding schedule and at the discretion of the Investigator.
- Total: Total of all reporting groups
Arm/Group | RAVICTI: Age 2 Months to < 2 Years | RAVICTI: Age 0 to <2 Months | Total
Number analyzed (Participants) | 10 | 16 | 26
Age, Continuous [Mean (Standard Deviation); unit: months] | 9.87 (5.529) | 0.83 (0.697) | 4.31 (5.606)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 7 | 12
  Male | 5 | 9 | 14

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Successful Transition to RAVICTI With Controlled Ammonia (i.e. No Clinical Symptoms and Ammonia < 100 μmol/L): Cohort of 2 Months to <2 Years Participants
Description: The percentage of participants with successful transition is based on Investigator response to the question, "Has transition to 100% RAVICTI been successful with controlled ammonia?" For participants 2 months of age and older, after a minimum of 24 hours of ammonia monitoring following the first full dose of RAVICTI alone, the participant was effectively transitioned when following conditions were met: no signs and symptoms of hyperammonemia; ammonia level less than 100 μmol/L (without normalization of ammonia, ie, without conversion of values from local laboratories with varying normal ranges to standardized values); and eligible for discharge per Investigator judgment.
Time Frame: Up to Day 4
Population: Safety Population: all enrolled participants who received any amount of study medication.
Measure: Number; unit: percentage of participants
Arm/Group | RAVICTI: Age 2 Months to < 2 Years
Number analyzed (Participants) | 10
percentage of participants | 100

2. Primary Outcome: Percentage of Participants With Successful Transition to RAVICTI With Controlled Ammonia (i.e. No Clinical Symptoms and Ammonia < 100 μmol/L): Cohort of 0 Months to <2 Months Participants
Description: The percentage of participants with successful transition is based on Investigator response to the question, "Has transition to 100% RAVICTI been successful with controlled ammonia?" For participants < 2 months of age, after a minimum of 24 hours of ammonia monitoring following the first full dose of RAVICTI alone, the participant was effectively transitioned when following conditions were met: no signs and symptoms of hyperammonemia; ammonia level less than 100 μmol/L (without normalization of ammonia, ie, without conversion of values from local laboratories with varying normal ranges to standardized values); and eligible for discharge per Investigator judgment.
Time Frame: Up to Day 4
Population: Safety Population: all enrolled participants who received any amount of study medication.
Measure: Number; unit: percentage of participants
Arm/Group | RAVICTI: Age 0 to < 2 Months
Number analyzed (Participants) | 16
percentage of participants | 100

3. Secondary Outcome: Rate of Hyperammonemic Crises (HACs): Cohort of 2 Months to <2 Years Participants
Description: HAC is defined having signs and symptoms consistent with hyperammonemia (such as but not limited to frequent vomiting, nausea, headache, lethargy, irritability, combativeness, and/or somnolence) associated with high blood ammonia and requiring medical intervention. Rate of HACs per 6 months during the safety extension is calculated as sum of (number of HAC) / sum of (days during first 6 months starting on Day 8 or number days on RAVICTI, whichever is less) across all participants in the corresponding group.
Time Frame: Day 8 through up to Month 6
Population: Safety Population: all enrolled participants who received any amount of study medication and had an assessment.
Measure: Number; unit: HACs per half-year of patient exposure
Arm/Group | RAVICTI: Age 2 Months to < 2 Years
Number analyzed (Participants) | 9
HACs per half-year of patient exposure | 0.005

4. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs), Serious TEAEs, Deaths, and Discontinuations Due to TEAEs: Cohort of 2 Months to <2 Years Participants
Description: An adverse event (AE) is any untoward medical occurrence, whether or not the event is considered related to the study drug. A serious AE is any AE that: results in death; is life threatening; requires hospitalization or prolongation of existing hospitalization; results in disability/incapacity; is a congenital anomaly/birth defect; is an important medical event. TEAEs are defined as AEs with an onset date on or after the first dose of study medication until study discontinuation. The Investigator assessed the causal relationship of each TEAE to the study drug as not related, possibly related, or probably related.
Time Frame: From the first dose of study treatment through 30 days after the final dose (mean [SD] duration of treatment was 9.13 [6.838] months).
Population: Safety Population: all enrolled participants who received any amount of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | RAVICTI: Age 2 Months to < 2 Years
Number analyzed (Participants) | 10
Participants
  ≥ 1 TEAE | 10
  ≥ 1 Related TEAE | 4
  ≥ 1 Serious TEAE | 6
  ≥ 1 Serious Related TEAE | 0
  Fatal Outcome TEAE | 1
  ≥ 1 TEAE Leading to Study Discontinuation | 1

5. Secondary Outcome: Amino Acid Assessment: Baseline and Change From Baseline in Glutamate Up to Month 24: Cohort of 2 Months to <2 Years Participants
Time Frame: Baseline, Day 7, Month 2, Month 3, Month 4, Month 5, Month 6, Month 9, Month 12, Month 15, Month 24
Population: Safety Population: all enrolled participants who received any amount of study medication and had an assessment at given time point.
Measure: Mean (Standard Deviation); unit: µmol/L
Arm/Group | RAVICTI: Age 2 Months to < 2 Years
Number analyzed (Participants) | 10
µmol/L
  Baseline: number analyzed (Participants) | 7
  Baseline | 122.43 (118.620)
  Day 7 change from Baseline: number analyzed (Participants) | 6
  Day 7 change from Baseline | -54.50 (92.626)
  Month 2 change from Baseline: number analyzed (Participants) | 5
  Month 2 change from Baseline | 7.80 (25.646)
  Month 3 change from Baseline: number analyzed (Participants) | 3
  Month 3 change from Baseline | -16.33 (39.209)
  Month 4 change from Baseline: number analyzed (Participants) | 4
  Month 4 change from Baseline | -13.00 (39.590)
  Month 5 change from Baseline: number analyzed (Participants) | 4
  Month 5 change from Baseline | 0.25 (13.426)
  Month 6 change from Baseline: number analyzed (Participants) | 5
  Month 6 change from Baseline | -2.20 (34.463)
  Month 9 change from Baseline: number analyzed (Participants) | 3
  Month 9 change from Baseline | 30.80 (17.092)
  Month 12 change from Baseline: number analyzed (Participants) | 3
  Month 12 change from Baseline | 22.20 (23.506)
  Month 15 change from Baseline: number analyzed (Participants) | 1
  Month 15 change from Baseline | 39.00 (NA) — 1 participant analyzed
  Month 24 change from Baseline: number analyzed (Participants) | 2
  Month 24 change from Baseline | 48.00 (53.740)

6. Secondary Outcome: Amino Acid Assessment: Baseline and Change From Baseline in Glutamine Up to Month 24: Cohort of 2 Months to <2 Years Participants
Time Frame: Baseline, Day 7, Month 2, Month 3, Month 4, Month 5, Month 6, Month 9, Month 12, Month 15, Month 24
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: µmol/L
Arm/Group | RAVICTI: Age 2 Months to < 2 Years
Number analyzed (Participants) | 10
µmol/L
  Baseline: number analyzed (Participants) | 7
  Baseline | 750.43 (309.000)
  Day 7 change from Baseline: number analyzed (Participants) | 6
  Day 7 change from Baseline | -184.33 (168.657)
  Month 2 change from Baseline: number analyzed (Participants) | 5
  Month 2 change from Baseline | -174.60 (318.249)
  Month 3 change from Baseline: number analyzed (Participants) | 3
  Month 3 change from Baseline | -374.00 (425.903)
  Month 4 change from Baseline: number analyzed (Participants) | 4
  Month 4 change from Baseline | -252.75 (323.852)
  Month 5 change from Baseline: number analyzed (Participants) | 4
  Month 5 change from Baseline | -370.25 (377.222)
  Month 6 change from Baseline: number analyzed (Participants) | 5
  Month 6 change from Baseline | -113.20 (519.710)
  Month 9 change from Baseline: number analyzed (Participants) | 3
  Month 9 change from Baseline | -446.53 (360.457)
  Month 12 change from Baseline: number analyzed (Participants) | 3
  Month 12 change from Baseline | -450.50 (386.699)
  Month 15 change from Baseline: number analyzed (Participants) | 1
  Month 15 change from Baseline | -149.00 (NA) — 1 participant with an assessment
  Month 24 change from Baseline: number analyzed (Participants) | 2
  Month 24 change from Baseline | 195.00 (554.372)

7. Secondary Outcome: Amino Acid Assessment: Baseline and Change From Baseline in Sum of Glutamine and Glutamate Up to Month 24: Cohort of 2 Months to <2 Years Participants
Time Frame: Baseline, Day 7, Month 2, Month 3, Month 4, Month 5, Month 6, Month 9, Month 12, Month 15, Month 24
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: µmol/L
Arm/Group | RAVICTI: Age 2 Months to < 2 Years
Number analyzed (Participants) | 10
µmol/L
  Baseline: number analyzed (Participants) | 7
  Baseline | 872.86 (381.005)
  Day 7 change from Baseline: number analyzed (Participants) | 6
  Day 7 change from Baseline | -238.83 (203.567)
  Month 2 change from Baseline: number analyzed (Participants) | 5
  Month 2 change from Baseline | -166.80 (332.421)
  Month 3 change from Baseline: number analyzed (Participants) | 3
  Month 3 change from Baseline | -390.33 (462.292)
  Month 4 change from Baseline: number analyzed (Participants) | 4
  Month 4 change from Baseline | -265.75 (339.015)
  Month 5 change from Baseline: number analyzed (Participants) | 4
  Month 5 change from Baseline | -370.00 (379.884)
  Month 6 change from Baseline: number analyzed (Participants) | 5
  Month 6 change from Baseline | -115.40 (546.796)
  Month 9 change from Baseline: number analyzed (Participants) | 3
  Month 9 change from Baseline | -415.73 (365.419)
  Month 12 change from Baseline: number analyzed (Participants) | 3
  Month 12 change from Baseline | -428.30 (404.351)
  Month 15 change from Baseline: number analyzed (Participants) | 1
  Month 15 change from Baseline | -110.00 (NA) — 1 participant with an assessment
  Month 24 change from Baseline: number analyzed (Participants) | 2
  Month 24 change from Baseline | 243.00 (608.112)

8. Secondary Outcome: Amino Acid Assessment: Baseline and Change From Baseline in Isoleucine Up to Month 24: Cohort of 2 Months to <2 Years Participants
Time Frame: Baseline, Day 7, Month 2, Month 3, Month 4, Month 5, Month 6, Month 9, Month 12, Month 15, Month 24
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: µmol/L
Arm/Group | RAVICTI: Age 2 Months to < 2 Years
Number analyzed (Participants) | 10
µmol/L
  Baseline: number analyzed (Participants) | 7
  Baseline | 54.86 (19.497)
  Day 7 change from Baseline: number analyzed (Participants) | 6
  Day 7 change from Baseline | 2.67 (19.159)
  Month 2 change from Baseline: number analyzed (Participants) | 5
  Month 2 change from Baseline | 4.20 (45.861)
  Month 3 change from Baseline: number analyzed (Participants) | 3
  Month 3 change from Baseline | -25.67 (16.743)
  Month 4 change from Baseline: number analyzed (Participants) | 4
  Month 4 change from Baseline | -20.25 (20.353)
  Month 5 change from Baseline: number analyzed (Participants) | 4
  Month 5 change from Baseline | -20.00 (36.341)
  Month 6 change from Baseline: number analyzed (Participants) | 5
  Month 6 change from Baseline | -16.40 (12.137)
  Month 9 change from Baseline: number analyzed (Participants) | 3
  Month 9 change from Baseline | -6.73 (13.342)
  Month 12 change from Baseline: number analyzed (Participants) | 3
  Month 12 change from Baseline | -13.33 (15.885)
  Month 15 change from Baseline: number analyzed (Participants) | 1
  Month 15 change from Baseline | -18.00 (NA) — 1 participant with an assessment
  Month 24 change from Baseline: number analyzed (Participants) | 2
  Month 24 change from Baseline | 1.50 (10.607)

9. Secondary Outcome: Amino Acid Assessment: Baseline and Change From Baseline in Leucine Up to Month 24: Cohort of 2 Months to <2 Years Participants
Time Frame: Baseline, Day 7, Month 2, Month 3, Month 4, Month 5, Month 6, Month 9, Month 12, Month 15, Month 24
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: µmol/L
Arm/Group | RAVICTI: Age 2 Months to < 2 Years
Number analyzed (Participants) | 10
µmol/L
  Baseline: number analyzed (Participants) | 7
  Baseline | 90.86 (29.249)
  Day 7 change from Baseline: number analyzed (Participants) | 6
  Day 7 change from Baseline | -0.83 (32.762)
  Month 2 change from Baseline: number analyzed (Participants) | 5
  Month 2 change from Baseline | 9.80 (65.975)
  Month 3 change from Baseline: number analyzed (Participants) | 3
  Month 3 change from Baseline | -33.00 (25.239)
  Month 4 change from Baseline: number analyzed (Participants) | 4
  Month 4 change from Baseline | -31.25 (24.771)
  Month 5 change from Baseline: number analyzed (Participants) | 4
  Month 5 change from Baseline | -39.50 (61.136)
  Month 6 change from Baseline: number analyzed (Participants) | 5
  Month 6 change from Baseline | -25.40 (13.594)
  Month 9 change from Baseline: number analyzed (Participants) | 3
  Month 9 change from Baseline | -19.13 (39.322)
  Month 12 change from Baseline: number analyzed (Participants) | 3
  Month 12 change from Baseline | -34.37 (23.283)
  Month 15 change from Baseline: number analyzed (Participants) | 1
  Month 15 change from Baseline | -40.00 (NA) — 1 participant with an assessment
  Month 24 change from Baseline: number analyzed (Participants) | 2
  Month 24 change from Baseline | -1.50 (31.820)

10. Secondary Outcome: Amino Acid Assessment: Baseline and Change From Baseline in Valine Up to Month 24: Cohort of 2 Months to <2 Years Participants
Time Frame: Baseline, Day 7, Month 2, Month 3, Month 4, Month 5, Month 6, Month 9, Month 12, Month 15, Month 24
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: µmol/L
Arm/Group | RAVICTI: Age 2 Months to < 2 Years
Number analyzed (Participants) | 10
µmol/L
  Baseline: number analyzed (Participants) | 7
  Baseline | 171.43 (42.887)
  Day 7 change from Baseline: number analyzed (Participants) | 6
  Day 7 change from Baseline | 4.00 (24.133)
  Month 2 change from Baseline: number analyzed (Participants) | 5
  Month 2 change from Baseline | 40.60 (90.057)
  Month 3 change from Baseline: number analyzed (Participants) | 3
  Month 3 change from Baseline | -27.33 (37.018)
  Month 4 change from Baseline: number analyzed (Participants) | 4
  Month 4 change from Baseline | -31.50 (29.760)
  Month 5 change from Baseline: number analyzed (Participants) | 4
  Month 5 change from Baseline | -56.00 (75.939)
  Month 6 change from Baseline: number analyzed (Participants) | 5
  Month 6 change from Baseline | -21.60 (18.202)
  Month 9 change from Baseline: number analyzed (Participants) | 3
  Month 9 change from Baseline | -11.90 (71.753)
  Month 12 change from Baseline: number analyzed (Participants) | 3
  Month 12 change from Baseline | -48.87 (51.644)
  Month 15 change from Baseline: number analyzed (Participants) | 1
  Month 15 change from Baseline | -46.00 (NA) — 1 participant with an assessment
  Month 24 change from Baseline: number analyzed (Participants) | 2
  Month 24 change from Baseline | 5.00 (55.154)

11. Secondary Outcome: Assessment of Growth and Development: Baseline and Change From Baseline in Body Mass Index (BMI) Z-Score Up to Month 24: Cohort of 2 Months to <2 Years Participants
Description: To assess any effect of study drug treatment on growth, Z-scores were calculated to express the deviation from a reference population for BMI. The Z-scores are based on the World Health Organization's Child Growth Standards charts. Negative Z-scores indicate lower than typical for age and gender while positive scores indicate higher than typical for age and gender.
Time Frame: Baseline, Month 1, Month 2, Month 3, Month 4, Month 5, Month 6, Month 9, Month 12, Month 15, Month 18, Month 24
Population: Safety Population: all enrolled participants who received any amount of study medication and had an assessment.
Measure: Mean (Standard Deviation); unit: z-score
Arm/Group | RAVICTI: Age 2 Months to < 2 Years
Number analyzed (Participants) | 10
z-score
  Baseline | 0.8107 (2.17017)
  Month 1 change from Baseline: number analyzed (Participants) | 9
  Month 1 change from Baseline | -0.2385 (0.77830)
  Month 2 change from Baseline: number analyzed (Participants) | 7
  Month 2 change from Baseline | -0.0249 (0.74861)
  Month 3 change from Baseline: number analyzed (Participants) | 7
  Month 3 change from Baseline | 0.1815 (0.86056)
  Month 4 change from Baseline: number analyzed (Participants) | 7
  Month 4 change from Baseline | 0.4434 (0.94854)
  Month 5 change from Baseline: number analyzed (Participants) | 6
  Month 5 change from Baseline | 0.1484 (0.76293)
  Month 6 change from Baseline: number analyzed (Participants) | 7
  Month 6 change from Baseline | 0.2497 (0.80923)
  Month 9 change from Baseline: number analyzed (Participants) | 5
  Month 9 change from Baseline | 0.6407 (0.98695)
  Month 12 change from Baseline: number analyzed (Participants) | 4
  Month 12 change from Baseline | 0.4164 (0.80674)
  Month 15 change from Baseline: number analyzed (Participants) | 2
  Month 15 change from Baseline | -0.2997 (0.16959)
  Month 18 change from Baseline: number analyzed (Participants) | 1
  Month 18 change from Baseline | -0.2038 (NA) — 1 participant with an assessment
  Month 24 change from Baseline: number analyzed (Participants) | 4
  Month 24 change from Baseline | 0.5581 (1.23993)

12. Secondary Outcome: Assessment of Growth and Development: Baseline and Change From Baseline in Body Surface Area (BSA) Z-Score Up to Month 24: Cohort of 2 Months to <2 Years Participants
Description: To assess any effect of study drug treatment on growth, Z-scores were calculated to express the deviation from a reference population for BSA. The Z-scores are based on weight-for-length charts. Negative Z-scores indicate lower than typical for age and gender while positive scores indicate higher than typical for age and gender.
Time Frame: Baseline, Month 1, Month 2, Month 3, Month 4, Month 5, Month 6, Month 9, Month 12, Month 15, Month 18, Month 24
Population: Safety Population: all enrolled participants who received any amount of study medication and had an assessment.
Measure: Mean (Standard Deviation); unit: z-score
Arm/Group | RAVICTI: Age 2 Months to < 2 Years
Number analyzed (Participants) | 10
z-score
  Baseline | 0.7143 (2.14922)
  Month 1 change from Baseline: number analyzed (Participants) | 9
  Month 1 change from Baseline | -0.2105 (0.74135)
  Month 2 change from Baseline: number analyzed (Participants) | 7
  Month 2 change from Baseline | -0.0704 (0.70393)
  Month 3 change from Baseline: number analyzed (Participants) | 7
  Month 3 change from Baseline | 0.1065 (0.70165)
  Month 4 change from Baseline: number analyzed (Participants) | 7
  Month 4 change from Baseline | 0.3365 (0.77672)
  Month 5 change from Baseline: number analyzed (Participants) | 6
  Month 5 change from Baseline | 0.1043 (0.56747)
  Month 6 change from Baseline: number analyzed (Participants) | 7
  Month 6 change from Baseline | 0.1842 (0.62205)
  Month 9 change from Baseline: number analyzed (Participants) | 5
  Month 9 change from Baseline | 0.4875 (0.86137)
  Month 12 change from Baseline: number analyzed (Participants) | 4
  Month 12 change from Baseline | 0.2944 (0.75133)
  Month 15 change from Baseline: number analyzed (Participants) | 2
  Month 15 change from Baseline | -0.3661 (0.00932)
  Month 18 change from Baseline: number analyzed (Participants) | 1
  Month 18 change from Baseline | -0.2214 (NA) — 1 participant with assessment
  Month 24 change from Baseline: number analyzed (Participants) | 4
  Month 24 change from Baseline | 0.4310 (1.13140)

13. Secondary Outcome: Plasma Phenylbutyrate/Phenylbutyric Acid (PBA) Maximum Plasma Concentration (Cmax) on the First Full Day of RAVICTI Dosing: Cohort of 2 Months to <2 Years Participants
Time Frame: Hour 0 and between 4 and 6 hours, 8 hours, and between 12 and 24 hours after the first dose of the day on Day 1 for stable participants and on Day 2 for participants in HAC
Population: Pharmacokinetic (PK) Evaluable Population: all participants from the safety population with individual concentration-time profiles that allow computation of meaningful PK parameter values.
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | RAVICTI: Age 2 Months to < 2 Years
Number analyzed (Participants) | 10
μg/mL | 42.44 (36.715)

14. Secondary Outcome: Plasma PBA Minimum Plasma Concentration (Cmin) on the First Full Day of RAVICTI Dosing: Cohort of 2 Months to <2 Years Participants
Time Frame: as for outcome 13
Population: PK Evaluable Population: all participants from the safety population with individual concentration-time profiles that allow computation of meaningful PK parameter values.
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | RAVICTI: Age 2 Months to < 2 Years
Number analyzed (Participants) | 10
μg/mL | 1.697 (2.254)

15. Secondary Outcome: Plasma PBA Area Under the Curve From Time Zero to the Time of Last Quantifiable Concentration (AUC[0-last]) on the First Full Day of RAVICTI Dosing: Cohort of 2 Months to <2 Years Participants
Time Frame: as for outcome 13
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: μg*hr/mL
Arm/Group | RAVICTI: Age 2 Months to < 2 Years
Number analyzed (Participants) | 10
μg*hr/mL | 280.936 (293.553)

16. Secondary Outcome: Plasma PBA Time to Cmax (Tmax) on the First Full Day of RAVICTI Dosing: Cohort of 2 Months to <2 Years Participants
Time Frame: as for outcome 13
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | RAVICTI: Age 2 Months to < 2 Years
Number analyzed (Participants) | 10
hours | 8.383 (4.564)

17. Secondary Outcome: Plasma Phenylacetate/Phenylacetic Acid (PAA) Cmax on the First Full Day of RAVICTI Dosing: Cohort of 2 Months to <2 Years Participants
Time Frame: as for outcome 13
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | RAVICTI: Age 2 Months to < 2 Years
Number analyzed (Participants) | 10
μg/mL | 36.52 (31.784)

18. Secondary Outcome: Plasma PAA Cmin on the First Full Day of RAVICTI Dosing: Cohort of 2 Months to <2 Years Participants
Time Frame: as for outcome 13
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | RAVICTI: Age 2 Months to < 2 Years
Number analyzed (Participants) | 10
μg/mL | 4.197 (6.434)

19. Secondary Outcome: Plasma PAA AUC(0-last) on the First Full Day of RAVICTI Dosing: Cohort of 2 Months to <2 Years Participants
Time Frame: as for outcome 13
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: μg*hr/mL
Arm/Group | RAVICTI: Age 2 Months to < 2 Years
Number analyzed (Participants) | 10
μg*hr/mL | 246.126 (238.547)

20. Secondary Outcome: Plasma PAA Tmax on the First Full Day of RAVICTI Dosing: Cohort of 2 Months to <2 Years Participants
Time Frame: as for outcome 13
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | RAVICTI: Age 2 Months to < 2 Years
Number analyzed (Participants) | 10
hours | 7.422 (7.351)

21. Secondary Outcome: Plasma Phenylacetylglutamine (PAGN) Cmax on the First Full Day of RAVICTI Dosing: Cohort of 2 Months to <2 Years Participants
Time Frame: as for outcome 13
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | RAVICTI: Age 2 Months to < 2 Years
Number analyzed (Participants) | 10
μg/mL | 62.45 (27.281)

22. Secondary Outcome: Plasma PAGN Cmin on the First Full Day of RAVICTI Dosing: Cohort of 2 Months to <2 Years Participants
Time Frame: as for outcome 13
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | RAVICTI: Age 2 Months to < 2 Years
Number analyzed (Participants) | 10
μg/mL | 20.62 (14.529)

23. Secondary Outcome: Plasma PAGN AUC(0-last) on the First Full Day of RAVICTI Dosing: Cohort of 2 Months to <2 Years Participants
Time Frame: as for outcome 13
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: μg*hr/mL
Arm/Group | RAVICTI: Age 2 Months to < 2 Years
Number analyzed (Participants) | 10
μg*hr/mL | 583.835 (285.241)

24. Secondary Outcome: Plasma PAGN Tmax on the First Full Day of RAVICTI Dosing: Cohort of 2 Months to <2 Years Participants
Time Frame: as for outcome 13
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | RAVICTI: Age 2 Months to < 2 Years
Number analyzed (Participants) | 10
hours | 6.573 (7.181)

25. Secondary Outcome: Assessment of Urinary PAGN Concentrations on the First Full Day of RAVICTI Dosing: Cohort of 2 Months to <2 Years Participants
Time Frame: Hour 0 and between 0.5 and 1 hour, 1.5 and 2.5 hours, 4 and 6 hours, 7.5 and 8.5 hours, and between 12 and 24 hours after the first dose of the day on Day 1 for stable participants and on Day 2 for participants in HAC
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | RAVICTI: Age 2 Months to < 2 Years
Number analyzed (Participants) | 10
μg/mL
  Hour 0: number analyzed (Participants) | 6
  Hour 0 | 3273 (1993)
  0.5 to 1.5 hours: number analyzed (Participants) | 6
  0.5 to 1.5 hours | 4140 (4399)
  1.5 to 2.5 hours: number analyzed (Participants) | 9
  1.5 to 2.5 hours | 3145 (5045)
  4 to 6 hours: number analyzed (Participants) | 9
  4 to 6 hours | 5202 (4547)
  7.5 to 8.5 hours: number analyzed (Participants) | 8
  7.5 to 8.5 hours | 3950 (3068)
  12 to 24 hours: number analyzed (Participants) | 9
  12 to 24 hours | 7561 (6956)

26. Secondary Outcome: Assessment of Urinary PAGN Concentrations Up to End of Trial: Cohort of 2 Months to <2 Years Participants
Time Frame: Day 7, Month 1, Month 2, Month 3, Month 4, Month 5, Month 6, Month 9, Month 12, Month 15, Month 18, End of Trial (up to Month 18)
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | RAVICTI: Age 2 Months to < 2 Years
Number analyzed (Participants) | 10
μg/mL
  Day 7: number analyzed (Participants) | 8
  Day 7 | 8859 (10500)
  Month 1: number analyzed (Participants) | 8
  Month 1 | 6274 (4802)
  Month 2: number analyzed (Participants) | 5
  Month 2 | 7386 (6419)
  Month 3: number analyzed (Participants) | 6
  Month 3 | 11456 (14471)
  Month 4: number analyzed (Participants) | 3
  Month 4 | 21416 (33695)
  Month 5: number analyzed (Participants) | 5
  Month 5 | 6129 (8024)
  Month 6: number analyzed (Participants) | 3
  Month 6 | 5347 (3153)
  Month 9: number analyzed (Participants) | 3
  Month 9 | 9357 (7286)
  Month 12: number analyzed (Participants) | 3
  Month 12 | 2580 (286)
  Month 15: number analyzed (Participants) | 1
  Month 15 | 6400 (NA) — 1 participant assessed
  Month 18: number analyzed (Participants) | 1
  Month 18 | 5250 (NA) — 1 participant assessed
  End of trial: number analyzed (Participants) | 3
  End of trial | 25333 (21324)

27. Secondary Outcome: Assessment of Urinary PAA Concentrations on the First Full Day of RAVICTI Dosing: Cohort of 2 Months to <2 Years Participants
Time Frame: Hour 0 and between 0.5 and 1.5 hours, 1.5 and 2.5 hours, 4 and 6 hours, 7.5 and 8.5 hours, and between 12 and 24 hours after the first dose of the day on Day 1 for stable participants and on Day 2 for participants in HAC
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | RAVICTI: Age 2 Months to < 2 Years
Number analyzed (Participants) | 10
μg/mL
  Hour 0: number analyzed (Participants) | 3
  Hour 0 | 18.78 (27.33)
  0.5 to 1.5 hours: number analyzed (Participants) | 4
  0.5 to 1.5 hours | 6.50 (3.39)
  1.5 to 2.5 hours: number analyzed (Participants) | 4
  1.5 to 2.5 hours | 7.29 (4.10)
  4 to 6 hours: number analyzed (Participants) | 6
  4 to 6 hours | 2.60 (2.18)
  7.5 to 8.5 hours: number analyzed (Participants) | 4
  7.5 to 8.5 hours | 4.48 (4.38)
  12 to 24 hours: number analyzed (Participants) | 4
  12 to 24 hours | 4.31 (2.33)

28. Secondary Outcome: Assessment of Urinary PAA Concentrations Up to End of Trial: Cohort of 2 Months to <2 Years Participants
Time Frame: Day 7, Month 1, Month 2, Month 3, Month 4, Month 5, Month 6, Month 9, Month 15, Month 18, End of Trial (up to Month 18)
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | RAVICTI: Age 2 Months to < 2 Years
Number analyzed (Participants) | 10
μg/mL
  Day 7: number analyzed (Participants) | 2
  Day 7 | 5.82 (2.21)
  Month 1: number analyzed (Participants) | 6
  Month 1 | 4.44 (4.61)
  Month 2: number analyzed (Participants) | 3
  Month 2 | 3.69 (1.82)
  Month 3: number analyzed (Participants) | 2
  Month 3 | 4.65 (0.49)
  Month 4: number analyzed (Participants) | 1
  Month 4 | 7.14 (NA) — 1 participant assessed
  Month 5: number analyzed (Participants) | 2
  Month 5 | 3.27 (1.96)
  Month 6: number analyzed (Participants) | 1
  Month 6 | 1.59 (NA) — 1 participant assessed
  Month 9: number analyzed (Participants) | 3
  Month 9 | 4.10 (1.65)
  Month 15: number analyzed (Participants) | 1
  Month 15 | 2.04 (NA) — 1 participant assessed
  Month 18: number analyzed (Participants) | 1
  Month 18 | 1.64 (NA) — 1 participant assessed
  End of trial: number analyzed (Participants) | 3
  End of trial | 7.0 (5.16)

29. Secondary Outcome: Rate of HACs: Cohort of 0 Months to <2 Months Participants
Description: HAC is defined as having signs and symptoms consistent with hyperammonemia (such as but not limited to frequent vomiting, nausea, headache, lethargy, irritability, combativeness, and/or somnolence) associated with high blood ammonia and requiring medical intervention. Rate of HACs per 6 months during the safety extension was calculated as sum of (number of HAC) / sum of (days during first 6 months starting on Day 8 or number days on RAVICTI, whichever is less) across all participants in the corresponding group.
Time Frame: Day 8 through up to Month 6
Population: Safety Population: all enrolled participants who received any amount of study medication.
Measure: Number; unit: HACs per half-year of patient exposure
Arm/Group | RAVICTI: Age 0 to < 2 Months
Number analyzed (Participants) | 16
HACs per half-year of patient exposure | 0.003

30. Secondary Outcome: Number of Participants With TEAEs, Serious TEAEs, Deaths, and Discontinuations Due to TEAEs: Cohort of 0 Months to <2 Months Participants
Description: An AE is any untoward medical occurrence, whether or not the event is considered related to the study drug. A serious AE is any AE that: results in death; is life threatening; requires hospitalization or prolongation of existing hospitalization; results in disability/incapacity; is a congenital anomaly/birth defect; is an important medical event. TEAEs are defined as AEs with an onset date on or after the first dose of study medication until study discontinuation. The Investigator assessed the causal relationship of each TEAE to the study drug as not related, possibly related, or probably related.
Time Frame: From the first dose of study treatment through 30 days after the final dose (mean [SD] duration of treatment was 10.67 [6.142] months).
Population: Safety Population: all enrolled participants who received any amount of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | RAVICTI: Age 0 to < 2 Months
Number analyzed (Participants) | 16
Participants
  ≥ 1 TEAE | 16
  ≥ 1 Related TEAE | 10
  ≥ 1 Serious TEAE | 11
  ≥ 1 Serious Related TEAE | 0
  Fatal Outcome TEAE | 0
  ≥ 1 TEAE Leading to Study Discontinuation | 1

31. Secondary Outcome: Amino Acid Assessment: Baseline and Change From Baseline in Glutamate Up to Month 24: Cohort of 0 Months to <2 Months Participants
Time Frame: Baseline, Day 7, Month 2, Month 3, Month 4, Month 5, Month 6, Month 9, Month 12, Month 15, Month 18, Month 24
Population: Safety Population: all enrolled participants who received any amount of study medication and had an assessment.
Measure: Mean (Standard Deviation); unit: μmol/L
Arm/Group | RAVICTI: Age 0 to < 2 Months
Number analyzed (Participants) | 16
μmol/L
  Baseline: number analyzed (Participants) | 15
  Baseline | 84.97 (52.086)
  Day 7 change from Baseline: number analyzed (Participants) | 14
  Day 7 change from Baseline | 26.81 (76.417)
  Month 2 change from Baseline: number analyzed (Participants) | 14
  Month 2 change from Baseline | 25.16 (64.474)
  Month 3 change from Baseline: number analyzed (Participants) | 14
  Month 3 change from Baseline | 50.05 (73.988)
  Month 4 change from Baseline: number analyzed (Participants) | 11
  Month 4 change from Baseline | 18.77 (67.561)
  Month 5 change from Baseline: number analyzed (Participants) | 10
  Month 5 change from Baseline | 57.43 (98.550)
  Month 6 change from Baseline: number analyzed (Participants) | 8
  Month 6 change from Baseline | 43.65 (140.985)
  Month 9 change from Baseline: number analyzed (Participants) | 8
  Month 9 change from Baseline | 33.41 (150.273)
  Month 12 change from Baseline: number analyzed (Participants) | 4
  Month 12 change from Baseline | 8.75 (97.329)
  Month 15 change from Baseline: number analyzed (Participants) | 4
  Month 15 change from Baseline | 25.75 (62.660)
  Month 18 change from Baseline: number analyzed (Participants) | 2
  Month 18 change from Baseline | 2.50 (21.920)
  Month 24 change from Baseline: number analyzed (Participants) | 8
  Month 24 change from Baseline | 16.10 (95.461)

32. Secondary Outcome: Amino Acid Assessment: Baseline and Change From Baseline in Glutamine Up to Month 24: Cohort of 0 Months to <2 Months Participants
Time Frame: Baseline, Day 7, Month 2, Month 3, Month 4, Month 5, Month 6, Month 9, Month 12, Month 15, Month 18, Month 24
Population: Safety Population: all enrolled participants who received any amount of study medication and had an assessment.
Measure: Mean (Standard Deviation); unit: μmol/L
Arm/Group | RAVICTI: Age 0 to < 2 Months
Number analyzed (Participants) | 16
μmol/L
  Baseline: number analyzed (Participants) | 15
  Baseline | 508.83 (337.175)
  Day 7 change from Baseline: number analyzed (Participants) | 14
  Day 7 change from Baseline | 21.04 (260.500)
  Month 2 change from Baseline: number analyzed (Participants) | 14
  Month 2 change from Baseline | -27.62 (379.796)
  Month 3 change from Baseline: number analyzed (Participants) | 14
  Month 3 change from Baseline | -15.09 (352.471)
  Month 4 change from Baseline: number analyzed (Participants) | 11
  Month 4 change from Baseline | -113.98 (230.855)
  Month 5 change from Baseline: number analyzed (Participants) | 10
  Month 5 change from Baseline | -99.82 (305.674)
  Month 6 change from Baseline: number analyzed (Participants) | 8
  Month 6 change from Baseline | -138.16 (349.269)
  Month 9 change from Baseline: number analyzed (Participants) | 8
  Month 9 change from Baseline | -56.08 (269.288)
  Month 12 change from Baseline: number analyzed (Participants) | 4
  Month 12 change from Baseline | -181.50 (118.604)
  Month 15 change from Baseline: number analyzed (Participants) | 4
  Month 15 change from Baseline | -103.75 (328.583)
  Month 18 change from Baseline: number analyzed (Participants) | 2
  Month 18 change from Baseline | -184.00 (80.610)
  Month 24 change from Baseline: number analyzed (Participants) | 8
  Month 24 change from Baseline | -219.93 (279.815)

33. Secondary Outcome: Amino Acid Assessment: Baseline and Change From Baseline in Sum of Glutamine and Glutamate Up to Month 24: Cohort of 0 Months to <2 Months Participants
Time Frame: Baseline, Day 7, Month 2, Month 3, Month 4, Month 5, Month 6, Month 9, Month 12, Month 15, Month 18, Month 24
Population: Safety Population: all enrolled participants who received any amount of study medication and had an assessment.
Measure: Mean (Standard Deviation); unit: μmol/L
Arm/Group | RAVICTI: Age 0 to < 2 Months
Number analyzed (Participants) | 16
μmol/L
  Baseline: number analyzed (Participants) | 15
  Baseline | 593.80 (333.657)
  Day 7 change from Baseline: number analyzed (Participants) | 14
  Day 7 change from Baseline | 47.85 (230.343)
  Month 2 change from Baseline: number analyzed (Participants) | 14
  Month 2 change from Baseline | -2.46 (402.919)
  Month 3 change from Baseline: number analyzed (Participants) | 14
  Month 3 change from Baseline | 34.96 (371.522)
  Month 4 change from Baseline: number analyzed (Participants) | 11
  Month 4 change from Baseline | -95.21 (238.136)
  Month 5 change from Baseline: number analyzed (Participants) | 10
  Month 5 change from Baseline | -42.39 (288.782)
  Month 6 change from Baseline: number analyzed (Participants) | 8
  Month 6 change from Baseline | -94.51 (297.378)
  Month 9 change from Baseline: number analyzed (Participants) | 8
  Month 9 change from Baseline | -22.66 (318.034)
  Month 12 change from Baseline: number analyzed (Participants) | 4
  Month 12 change from Baseline | -172.75 (210.202)
  Month 15 change from Baseline: number analyzed (Participants) | 4
  Month 15 change from Baseline | -78.00 (297.410)
  Month 18 change from Baseline: number analyzed (Participants) | 2
  Month 18 change from Baseline | -181.50 (102.530)
  Month 24 change from Baseline: number analyzed (Participants) | 8
  Month 24 change from Baseline | -203.83 (255.810)

34. Secondary Outcome: Amino Acid Assessment: Baseline and Change From Baseline in Isoleucine Up to Month 24: Cohort of 0 Months to <2 Months Participants
Time Frame: Baseline, Day 7, Month 2, Month 3, Month 4, Month 5, Month 6, Month 9, Month 12, Month 15, Month 18, Month 24
Population: Safety Population: all enrolled participants who received any amount of study medication and had an assessment.
Measure: Mean (Standard Deviation); unit: μmol/L
Arm/Group | RAVICTI: Age 0 to < 2 Months
Number analyzed (Participants) | 16
μmol/L
  Baseline: number analyzed (Participants) | 15
  Baseline | 142.68 (222.694)
  Day 7 change from Baseline: number analyzed (Participants) | 14
  Day 7 change from Baseline | -49.09 (198.730)
  Month 2 change from Baseline: number analyzed (Participants) | 14
  Month 2 change from Baseline | -1.62 (233.754)
  Month 3 change from Baseline: number analyzed (Participants) | 14
  Month 3 change from Baseline | -20.46 (216.885)
  Month 4 change from Baseline: number analyzed (Participants) | 11
  Month 4 change from Baseline | -67.32 (173.564)
  Month 5 change from Baseline: number analyzed (Participants) | 10
  Month 5 change from Baseline | -75.45 (221.845)
  Month 6 change from Baseline: number analyzed (Participants) | 8
  Month 6 change from Baseline | -35.94 (78.367)
  Month 9 change from Baseline: number analyzed (Participants) | 8
  Month 9 change from Baseline | -73.09 (245.051)
  Month 12 change from Baseline: number analyzed (Participants) | 4
  Month 12 change from Baseline | -178.50 (335.538)
  Month 15 change from Baseline: number analyzed (Participants) | 4
  Month 15 change from Baseline | -139.50 (359.287)
  Month 18 change from Baseline: number analyzed (Participants) | 2
  Month 18 change from Baseline | 1.00 (45.255)
  Month 24 change from Baseline: number analyzed (Participants) | 8
  Month 24 change from Baseline | -55.31 (217.209)

35. Secondary Outcome: Amino Acid Assessment: Baseline and Change From Baseline in Leucine Up to Month 24: Cohort of 0 Months to <2 Months Participants
Time Frame: Baseline, Day 7, Month 2, Month 3, Month 4, Month 5, Month 6, Month 9, Month 12, Month 15, Month 18, Month 24
Population: Safety Population: all enrolled participants who received any amount of study medication and had an assessment.
Measure: Mean (Standard Deviation); unit: μmol/L
Arm/Group | RAVICTI: Age 0 to < 2 Months
Number analyzed (Participants) | 16
μmol/L
  Baseline: number analyzed (Participants) | 15
  Baseline | 133.67 (253.829)
  Day 7 change from Baseline: number analyzed (Participants) | 14
  Day 7 change from Baseline | -81.91 (273.127)
  Month 2 change from Baseline: number analyzed (Participants) | 14
  Month 2 change from Baseline | -60.80 (278.083)
  Month 3 change from Baseline: number analyzed (Participants) | 14
  Month 3 change from Baseline | -51.66 (269.558)
  Month 4 change from Baseline: number analyzed (Participants) | 11
  Month 4 change from Baseline | -82.82 (224.269)
  Month 5 change from Baseline: number analyzed (Participants) | 10
  Month 5 change from Baseline | -118.55 (311.125)
  Month 6 change from Baseline: number analyzed (Participants) | 8
  Month 6 change from Baseline | -11.85 (40.693)
  Month 9 change from Baseline: number analyzed (Participants) | 8
  Month 9 change from Baseline | -115.09 (338.186)
  Month 12 change from Baseline: number analyzed (Participants) | 4
  Month 12 change from Baseline | -249.50 (483.776)
  Month 15 change from Baseline: number analyzed (Participants) | 4
  Month 15 change from Baseline | -195.75 (496.313)
  Month 18 change from Baseline: number analyzed (Participants) | 2
  Month 18 change from Baseline | 6.00 (62.225)
  Month 24 change from Baseline: number analyzed (Participants) | 8
  Month 24 change from Baseline | -82.54 (228.107)

36. Secondary Outcome: Amino Acid Assessment: Baseline and Change From Baseline in Valine Up to Month 24: Cohort of 0 Months to <2 Months Participants
Time Frame: Baseline, Day 7, Month 2, Month 3, Month 4, Month 5, Month 6, Month 9, Month 12, Month 15, Month 18, Month 24
Population: Safety Population: all enrolled participants who received any amount of study medication and had an assessment.
Measure: Mean (Standard Deviation); unit: μmol/L
Arm/Group | RAVICTI: Age 0 to < 2 Months
Number analyzed (Participants) | 16
μmol/L
  Baseline: number analyzed (Participants) | 15
  Baseline | 181.49 (257.948)
  Day 7 change from Baseline: number analyzed (Participants) | 14
  Day 7 change from Baseline | -63.96 (290.312)
  Month 2 change from Baseline: number analyzed (Participants) | 14
  Month 2 change from Baseline | -39.04 (297.634)
  Month 3 change from Baseline: number analyzed (Participants) | 14
  Month 3 change from Baseline | -23.86 (290.128)
  Month 4 change from Baseline: number analyzed (Participants) | 11
  Month 4 change from Baseline | -74.41 (233.538)
  Month 5 change from Baseline: number analyzed (Participants) | 10
  Month 5 change from Baseline | -98.67 (326.300)
  Month 6 change from Baseline: number analyzed (Participants) | 8
  Month 6 change from Baseline | 2.64 (77.843)
  Month 9 change from Baseline: number analyzed (Participants) | 8
  Month 9 change from Baseline | -90.40 (355.316)
  Month 12 change from Baseline: number analyzed (Participants) | 4
  Month 12 change from Baseline | -238.25 (506.435)
  Month 15 change from Baseline: number analyzed (Participants) | 4
  Month 15 change from Baseline | -137.00 (519.042)
  Month 18 change from Baseline: number analyzed (Participants) | 2
  Month 18 change from Baseline | 38.00 (67.882)
  Month 24 change from Baseline: number analyzed (Participants) | 8
  Month 24 change from Baseline | -72.78 (258.710)

37. Secondary Outcome: Assessment of Growth and Development: Baseline and Change From Baseline in BMI Z-Score Up to Month 24: Cohort of 0 Months to <2 Months Participants
Description: as for outcome 11
Time Frame: Baseline, Month 1, Month 2, Month 3, Month 4, Month 5, Month 6, Month 9, Month 12, Month 15, Month 18, Month 24
Population: Safety Population: all enrolled participants who received any amount of study medication and had an assessment.
Measure: Mean (Standard Deviation); unit: z-score
Arm/Group | RAVICTI: Age 0 to < 2 Months
Number analyzed (Participants) | 16
z-score
  Baseline | -0.0544 (1.26821)
  Month 1 change from Baseline | -0.2158 (1.35960)
  Month 2 change from Baseline: number analyzed (Participants) | 15
  Month 2 change from Baseline | -0.2598 (1.19544)
  Month 3 change from Baseline: number analyzed (Participants) | 15
  Month 3 change from Baseline | -0.1617 (1.02572)
  Month 4 change from Baseline: number analyzed (Participants) | 12
  Month 4 change from Baseline | -0.0264 (1.68215)
  Month 5 change from Baseline: number analyzed (Participants) | 11
  Month 5 change from Baseline | 0.0828 (1.14206)
  Month 6 change from Baseline: number analyzed (Participants) | 10
  Month 6 change from Baseline | 0.0136 (1.72106)
  Month 9 change from Baseline: number analyzed (Participants) | 9
  Month 9 change from Baseline | 0.4614 (1.25343)
  Month 12 change from Baseline: number analyzed (Participants) | 6
  Month 12 change from Baseline | 0.6646 (0.95334)
  Month 15 change from Baseline: number analyzed (Participants) | 4
  Month 15 change from Baseline | 0.6830 (0.55703)
  Month 18 change from Baseline: number analyzed (Participants) | 3
  Month 18 change from Baseline | 0.3308 (0.27572)
  Month 24 change from Baseline: number analyzed (Participants) | 10
  Month 24 change from Baseline | 0.7743 (0.64962)

38. Secondary Outcome: Assessment of Growth and Development: Baseline and Change From Baseline in BSA Z-Score Up to Month 24: Cohort of 0 Months to <2 Months Participants
Description: as for outcome 12
Time Frame: Baseline, Month 1, Month 2, Month 3, Month 4, Month 5, Month 6, Month 9, Month 12, Month 15, Month 18, Month 24
Population: Safety Population: all enrolled participants who received any amount of study medication and had an assessment.
Measure: Mean (Standard Deviation); unit: z-score
Arm/Group | RAVICTI: Age 0 to < 2 Months
Number analyzed (Participants) | 16
z-score
  Baseline | -0.1980 (2.11774)
  Month 1 change from Baseline | 0.2336 (1.95603)
  Month 2 change from Baseline: number analyzed (Participants) | 15
  Month 2 change from Baseline | 0.2006 (1.72135)
  Month 3 change from Baseline: number analyzed (Participants) | 15
  Month 3 change from Baseline | 0.2684 (1.37517)
  Month 4 change from Baseline: number analyzed (Participants) | 12
  Month 4 change from Baseline | 0.2372 (2.30831)
  Month 5 change from Baseline: number analyzed (Participants) | 11
  Month 5 change from Baseline | 0.1810 (1.70024)
  Month 6 change from Baseline: number analyzed (Participants) | 10
  Month 6 change from Baseline | 0.2902 (2.05956)
  Month 9 change from Baseline: number analyzed (Participants) | 9
  Month 9 change from Baseline | 0.1679 (1.32407)
  Month 12 change from Baseline: number analyzed (Participants) | 6
  Month 12 change from Baseline | 0.1308 (0.50371)
  Month 15 change from Baseline: number analyzed (Participants) | 4
  Month 15 change from Baseline | 0.1595 (0.75833)
  Month 18 change from Baseline: number analyzed (Participants) | 3
  Month 18 change from Baseline | 0.1050 (0.73521)
  Month 24 change from Baseline: number analyzed (Participants) | 10
  Month 24 change from Baseline | 0.7341 (1.35582)

39. Secondary Outcome: Plasma PBA Cmax on the First Full Day of RAVICTI Dosing: Cohort of 0 Months to <2 Months Participants
Time Frame: as for outcome 13
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | RAVICTI: Age 0 to < 2 Months
Number analyzed (Participants) | 16
μg/mL | 46.2 (49.8)

40. Secondary Outcome: Plasma PBA Cmin on the First Full Day of RAVICTI Dosing: Cohort of 0 Months to <2 Months Participants
Time Frame: as for outcome 13
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | RAVICTI: Age 0 to < 2 Months
Number analyzed (Participants) | 7
μg/mL | 4.8 (4.2)

41. Secondary Outcome: Plasma PBA AUC(0-last) on the First Full Day of RAVICTI Dosing: Cohort of 0 Months to <2 Months Participants
Time Frame: as for outcome 13
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: μg*hr/mL
Arm/Group | RAVICTI: Age 0 to < 2 Months
Number analyzed (Participants) | 16
μg*hr/mL | 374.53 (390.48)

42. Secondary Outcome: Plasma PBA Tmax on the First Full Day of RAVICTI Dosing: Cohort of 0 Months to <2 Months Participants
Time Frame: as for outcome 13
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | RAVICTI: Age 0 to < 2 Months
Number analyzed (Participants) | 16
hours | 9.39 (7.41)

43. Secondary Outcome: Plasma PAA Cmax on the First Full Day of RAVICTI Dosing: Cohort of 0 Months to <2 Months Participants
Time Frame: as for outcome 13
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | RAVICTI: Age 0 to < 2 Months
Number analyzed (Participants) | 16
μg/mL | 115.3 (102.0)

44. Secondary Outcome: Plasma PAA Cmin on the First Full Day of RAVICTI Dosing: Cohort of 0 Months to <2 Months Participants
Time Frame: as for outcome 13
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | RAVICTI: Age 0 to < 2 Months
Number analyzed (Participants) | 10
μg/mL | 98.98 (122.07)

45. Secondary Outcome: Plasma PAA AUC(0-last) on the First Full Day of RAVICTI Dosing: Cohort of 0 Months to <2 Months Participants
Time Frame: as for outcome 13
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: μg*hr/mL
Arm/Group | RAVICTI: Age 0 to < 2 Months
Number analyzed (Participants) | 16
μg*hr/mL | 1321.18 (1220.52)

46. Secondary Outcome: Plasma PAA Tmax on the First Full Day of RAVICTI Dosing: Cohort of 0 Months to <2 Months Participants
Time Frame: as for outcome 13
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | RAVICTI: Age 0 to < 2 Months
Number analyzed (Participants) | 16
hours | 9.85 (9.26)

47. Secondary Outcome: Plasma PAGN Cmax on the First Full Day of RAVICTI Dosing: Cohort of 0 Months to <2 Months Participants
Time Frame: as for outcome 13
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | RAVICTI: Age 0 to < 2 Months
Number analyzed (Participants) | 16
μg/mL | 102.1 (48.6)

48. Secondary Outcome: Plasma PAGN Cmin on the First Full Day of RAVICTI Dosing: Cohort of 0 Months to <2 Months Participants
Time Frame: as for outcome 13
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | RAVICTI: Age 0 to < 2 Months
Number analyzed (Participants) | 13
μg/mL | 69.39 (54.03)

49. Secondary Outcome: Plasma PAGN AUC(0-last) on the First Full Day of RAVICTI Dosing: Cohort of 0 Months to <2 Months Participants
Time Frame: as for outcome 13
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: μg*hr/mL
Arm/Group | RAVICTI: Age 0 to < 2 Months
Number analyzed (Participants) | 16
μg*hr/mL | 1384.12 (1141.03)

50. Secondary Outcome: Plasma PAGN Tmax on the First Full Day of RAVICTI Dosing: Cohort of 0 Months to <2 Months Participants
Time Frame: as for outcome 13
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | RAVICTI: Age 0 to < 2 Months
Number analyzed (Participants) | 16
hours | 11.72 (8.24)

51. Secondary Outcome: Assessment of Urinary PAGN Concentrations on the First Full Day of RAVICTI Dosing: Cohort of 0 Months to <2 Months Participants
Time Frame: as for outcome 25
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | RAVICTI: Age 0 to < 2 Months
Number analyzed (Participants) | 16
μg/mL
  Hour 0: number analyzed (Participants) | 6
  Hour 0 | 3530.43 (3600.4)
  0.5 to 1.5 hours: number analyzed (Participants) | 8
  0.5 to 1.5 hours | 1828 (2862)
  1.5 to 2.5 hours: number analyzed (Participants) | 9
  1.5 to 2.5 hours | 1746 (1464)
  4 to 6 hours: number analyzed (Participants) | 11
  4 to 6 hours | 2260 (1472)
  7.5 to 8.5 hours: number analyzed (Participants) | 14
  7.5 to 8.5 hours | 3530.43 (3600.4)
  12 to 24 hours | 4404 (3766)

52. Secondary Outcome: Assessment of Urinary PAGN Concentrations Up to End of Trial: Cohort of 0 Months to <2 Months Participants
Time Frame: Day 7, Month 1, Month 2, Month 3, Month 4, Month 5, Month 6, Month 9, Month 12, Month 15, End of Trial (up to Month 15)
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | RAVICTI: Age 0 to < 2 Months
Number analyzed (Participants) | 16
μg/mL
  Day 7: number analyzed (Participants) | 10
  Day 7 | 4643 (2506)
  Month 1: number analyzed (Participants) | 11
  Month 1 | 4517 (2485)
  Month 2: number analyzed (Participants) | 12
  Month 2 | 4116 (3137)
  Month 3: number analyzed (Participants) | 9
  Month 3 | 7037 (4493)
  Month 4: number analyzed (Participants) | 9
  Month 4 | 2826 (1543)
  Month 5: number analyzed (Participants) | 8
  Month 5 | 6973 (3682)
  Month 6: number analyzed (Participants) | 3
  Month 6 | 5883 (3128)
  Month 9: number analyzed (Participants) | 7
  Month 9 | 7006 (4289)
  Month 12: number analyzed (Participants) | 3
  Month 12 | 5847 (2992)
  Month 15: number analyzed (Participants) | 4
  Month 15 | 3915 (2584)
  End of trial: number analyzed (Participants) | 8
  End of trial | 6939 (6581)

53. Secondary Outcome: Assessment of Urinary PAA Concentrations on the First Full Day of RAVICTI Dosing: Cohort of 0 Months to <2 Months Participants
Time Frame: as for outcome 27
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | RAVICTI: Age 0 to < 2 Months
Number analyzed (Participants) | 16
μg/mL
  Hour 0: number analyzed (Participants) | 3
  Hour 0 | 11.1 (10.4)
  0.5 to 1.5 hours: number analyzed (Participants) | 4
  0.5 to 1.5 hours | 46.2 (58.6)
  1.5 to 2.5 hours: number analyzed (Participants) | 4
  1.5 to 2.5 hours | 62.5 (42.8)
  4 to 6 hours: number analyzed (Participants) | 9
  4 to 6 hours | 34.6 (56.2)
  7.5 to 8.5 hours: number analyzed (Participants) | 11
  7.5 to 8.5 hours | 22.8 (25.3)
  12 to 24 hours: number analyzed (Participants) | 12
  12 to 24 hours | 35.2 (51.0)

54. Secondary Outcome: Assessment of Urinary PAA Concentrations Up to End of Trial: Cohort of 0 Months to <2 Months Participants
Time Frame: Day 7, Month 1, Month 2, Month 3, Month 4, Month 5, Month 6, Month 9, Month 15, End of Trial (up to Month 15)
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | RAVICTI: Age 0 to < 2 Months
Number analyzed (Participants) | 16
μg/mL
  Day 7: number analyzed (Participants) | 9
  Day 7 | 23.7 (31.2)
  Month 1: number analyzed (Participants) | 8
  Month 1 | 14.6 (17.2)
  Month 2: number analyzed (Participants) | 8
  Month 2 | 12.3 (13.3)
  Month 3: number analyzed (Participants) | 7
  Month 3 | 14.4 (10.7)
  Month 4: number analyzed (Participants) | 6
  Month 4 | 6.4 (7.1)
  Month 5: number analyzed (Participants) | 6
  Month 5 | 13.2 (14.0)
  Month 6: number analyzed (Participants) | 1
  Month 6 | 5.5 (NA) — 1 participant assessed
  Month 9: number analyzed (Participants) | 7
  Month 9 | 11.8 (8.5)
  Month 12: number analyzed (Participants) | 3
  Month 12 | 6.0 (3.8)
  Month 15: number analyzed (Participants) | 2
  Month 15 | 4.9 (0.3)
  End of trial: number analyzed (Participants) | 5
  End of trial | 11.6 (9.0)

ADVERSE EVENTS:
Time Frame: From the first dose of study treatment through 30 days after the final dose (mean [SD] duration of treatment was 9.13 [6.838] months for Cohort of 2 Months to <2 Years Participants and 10.67 [6.142] months for Cohort of 0 Months to <2 Months Participants).
Description: TEAEs (defined as AEs with an onset date on or after the first dose of study medication until study discontinuation) are presented.
Arm/Group | RAVICTI: Age 2 Months to < 2 Years | RAVICTI: Age 0 to <2 Months
All-Cause Mortality (participants affected / at risk) | 1/10 | 0/16
Serious Adverse Events (participants affected / at risk) | 6/10 | 11/16
Other Adverse Events (participants affected / at risk) | 8/10 | 16/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | RAVICTI: Age 2 Months to < 2 Years (N=10) | RAVICTI: Age 0 to <2 Months (N=16)
Ammonia increased (Investigations) | 1 | 0
Cyanosis (Cardiac disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 1
Apnoeic attack (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Status asthmaticus (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Lethargy (Nervous system disorders) | 0 | 1
Pyrexia (General disorders) | 1 | 0
Pneumatosis intestinalis (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 2
Hyperammonaemia (Metabolism and nutrition disorders) | 3 | 5
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Feeding disorder (Metabolism and nutrition disorders) | 0 | 1
Croup infectious (Infections and infestations) | 1 | 1
Gastroenteritis (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 1
Viral infection (Infections and infestations) | 2 | 1
Influenza (Infections and infestations) | 1 | 0
Peritonitis (Infections and infestations) | 1 | 0
Rhinovirus infection (Infections and infestations) | 1 | 0
Viral upper respiratory tract infection (Infections and infestations) | 1 | 0
Bacteraemia (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 0 | 1
Device related infection (Infections and infestations) | 0 | 1
Medical device site infection (Infections and infestations) | 0 | 1
Meningitis bacterial (Infections and infestations) | 0 | 1
Respiratory syncytial virus infection (Infections and infestations) | 0 | 1
Tracheitis (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | RAVICTI: Age 2 Months to < 2 Years (N=10) | RAVICTI: Age 0 to <2 Months (N=16)
Venous thrombosis limb (Vascular disorders) | 1 | 0
Seasonal allergy (Immune system disorders) | 1 | 0
Pyrexia (General disorders) | 2 | 2
Catheter site rash (General disorders) | 0 | 1
Device occlusion (General disorders) | 0 | 1
Drug withdrawal syndrome (General disorders) | 0 | 1
Medical device site haemorrhage (General disorders) | 0 | 1
Agitation (Psychiatric disorders) | 0 | 1
Irritability (Psychiatric disorders) | 0 | 1
Stoma site reaction (Injury, poisoning and procedural complications) | 1 | 1
Tibia fracture (Injury, poisoning and procedural complications) | 1 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 1
Amino acid level decreased (Investigations) | 1 | 1
Ammonia increased (Investigations) | 1 | 1
Carbon dioxide decreased (Investigations) | 1 | 1
Hepatic enzyme increased (Investigations) | 0 | 2
Alanine aminotransferase increased (Investigations) | 0 | 1
Amino acid level increased (Investigations) | 0 | 1
Anion gap increased (Investigations) | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 1
Blood bicarbonate decreased (Investigations) | 0 | 1
Blood urea decreased (Investigations) | 0 | 1
Body height below normal (Investigations) | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 0 | 1
Platelet count increased (Investigations) | 0 | 1
Transaminases increased (Investigations) | 0 | 1
Weight decreased (Investigations) | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 1
Dacryostenosis congenital (Congenital, familial and genetic disorders) | 1 | 0
Plagiocephaly (Congenital, familial and genetic disorders) | 0 | 2
Anaemia (Blood and lymphatic system disorders) | 1 | 3
Neutropenia (Blood and lymphatic system disorders) | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 2
Thrombocytosis (Blood and lymphatic system disorders) | 0 | 2
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1
Lymphocytosis (Blood and lymphatic system disorders) | 0 | 1
Microcytic anaemia (Blood and lymphatic system disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 4
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Apnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Use of accessory respiratory muscles (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Gross motor delay (Nervous system disorders) | 1 | 0
Lethargy (Nervous system disorders) | 0 | 1
Tremor (Nervous system disorders) | 0 | 1
Eye discharge (Eye disorders) | 0 | 1
Ocular hyperaemia (Eye disorders) | 0 | 1
Excessive cerumen production (Ear and labyrinth disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 5
Vomiting (Gastrointestinal disorders) | 4 | 5
Teething (Gastrointestinal disorders) | 1 | 3
Constipation (Gastrointestinal disorders) | 2 | 2
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 6
Flatulence (Gastrointestinal disorders) | 0 | 3
Dysphagia (Gastrointestinal disorders) | 0 | 1
Post-tussive vomiting (Gastrointestinal disorders) | 0 | 1
Hepatic calcification (Hepatobiliary disorders) | 0 | 1
Vesicoureteric reflux (Renal and urinary disorders) | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 1
Nail ridging (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 5
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 1 | 6
Eczema (Skin and subcutaneous tissue disorders) | 1 | 1
Red man syndrome (Skin and subcutaneous tissue disorders) | 0 | 1
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1
Torticollis (Musculoskeletal and connective tissue disorders) | 0 | 1
Metabolic acidosis (Metabolism and nutrition disorders) | 2 | 2
Hypophagia (Metabolism and nutrition disorders) | 2 | 1
Hyperammonaemia (Metabolism and nutrition disorders) | 0 | 2
Dehydration (Metabolism and nutrition disorders) | 0 | 2
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1
Feeding disorder of infancy or early childhood (Metabolism and nutrition disorders) | 0 | 1
Protein deficiency (Metabolism and nutrition disorders) | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 1
Upper respiratory tract infection (Infections and infestations) | 4 | 5
Urinary tract infection (Infections and infestations) | 1 | 2
Viral infection (Infections and infestations) | 1 | 1
Nasopharyngitis (Infections and infestations) | 2 | 4
Croup infectious (Infections and infestations) | 1 | 1
Otitis media (Infections and infestations) | 2 | 1
Conjunctivitis (Infections and infestations) | 1 | 0
Pharyngitis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0
Sinusitis (Infections and infestations) | 1 | 1
Ear infection (Infections and infestations) | 0 | 3
Oral candidiasis (Infections and infestations) | 0 | 2
Respiratory syncytial virus infection (Infections and infestations) | 0 | 1
Angular cheilitis (Infections and infestations) | 0 | 1
Candida infection (Infections and infestations) | 0 | 1
Gastrointestinal viral infection (Infections and infestations) | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 1
Otitis media acute (Infections and infestations) | 0 | 1
Rhinovirus infection (Infections and infestations) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Horizon requests that any investigator/institution that plans on presenting/publishing results provide written notification of their request 60 days prior to their presentation/publication. Horizon requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if Horizon needs to secure patent or proprietary protection.